CLINICAL TRIAL: NCT02422316
Title: Non-contrast Cardiac CT as a Risk Stratification Tool in Patients With Non-cardiac Chest Pain
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, associate professor, University of Southern Denmark
Other Study IDs: SHS-ED-2014-01
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-contrast Cardiac CT scan

SUMMARY:
Background:

Only around 20% of all patients seen in hospital with suspected Acute Coronary Syndrome will have Acute Myocardial Infarction. However, several studies indicate that patients where ACS had been excluded by conventional methods sustain a higher cardiac morbidity and mortality than the background population. Not all of these patients can be identified by traditional risk factors such as cholesterol, hypertension, and diabetes or with conventional methods such as ECG, troponin and clinical symptoms. Non-Contrast Cardiac-CT measures the amount of calcification in the coronary arteries and might be a useful addition in predicting future cardiac events in this patient group. The aim of this study is through a double-blinded study to determine whether non-contrast CT scan with calcium score can be used to identify patients at increased risk of death and cardiac event within the following 12 months after an acute admission where troponin measurements were normal.

Methods:

The study will investigate patients with suspected Acute Coronary syndrome who have been examined and subsequently sent home from an emergency- or cardiology department without ACS or another obvious explanation. 750 patients, age 30-70 years who are included in the study: "Identification of risk factors in non-cardiac chest pain patients" will be offered a non-contrast CT scan with calcium score within 14 days after the hospital contact. The participants will be included in a 12 months follow up, where the result of the calcium score is not revealed neither for the patient nor the investigator. After 12 months the results of the scan is compared with the rate of cardiac events. This project is a multicenter study and recruits patients from 6 emergency - and cardiology departments in the region of Southern Denmark.

The study commences at September 2014 and results of this project are expected to contribute to the risk stratification of Non-cardiac chest pain patients.

ELIGIBILITY:
Inclusion Criteria:

* chest pain with normal cardiac enzymes.
* legal competent
* age 30-70 years

Exclusion Criteria:

* chest pain of obvious reason
* previous acute coronary syndrome
* previous coronary artery investigations within last five years
* patients referred for other cardiac examinations after the current admission

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will investigate patients with suspected Acute Coronary syndrome who have been examined and subsequently sent home from an emergency- or cardiology department without ACS or another obvious explanation. 750 patients, age 30-70 years
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
major cardiac events | one year
  major cardiac events: cardiac deaths, revascularization, ischaemic related arrythmias, cardiac related readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Aabenraa, Denmark

REFERENCES:
- [Derived] Ilangkovan N, Mogensen CB, Mickley H, Lassen AT, Lambrechtsen J, Sand NPR, Albiniussen R, Byg J, Steffensen FH, Gronhoj MH, Diederichsen A. Prevalence of coronary artery calcification in a non-specific chest pain population in emergency and cardiology departments compared with the background population: a prospective cohort study in Southern Denmark with 12-month follow-up of cardiac endpoints. BMJ Open. 2018 Mar 3;8(3):e018391. doi: 10.1136/bmjopen-2017-018391. PMID 29502085